CLINICAL TRIAL: NCT05087784
Title: AlloLife - Life After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: AlloLife - Life After Transplantation
Acronym: AlloLife
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Collaborators: Universität des Saarlandes (Other); Institut Paoli-Calmettes (Other); Medical University of Warsaw (Other); University Of Perugia (Other); Centre for Research and Technology Hellas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20210920H
Record Dates: First submitted 2021-09-20; First posted 2021-10-21 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Survivorship; Stem Cell Transplant Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: (Experimental): Complex, technology supported survivorship intervention using wearable devices for patients, supportive patient apps and physician apps for risk prediction. Increased Cardio-oncology visits assigned to risk patients as predicted by the app.
  Interventions: Combination Product: Technology supported, coordinated survivorship care using wearable devices, supportive patient-apps and cardio-oncology physician apps
- Control arm: (No Intervention): Wearable device for patients together with a basic patient app providing feedback on the wearable device records and patient information material.

INTERVENTIONS:
Combination Product: Technology supported, coordinated survivorship care using wearable devices, supportive patient-apps and cardio-oncology physician apps — Patient-centered, technology-supported integrated survivorship- and care management
  Arms: Intervention:

SUMMARY:
Survivors of allo HCT can experience long-term survival, which is however limited by a number of late effects. These will be addressed in AlloLife to improve quality of life (QoL) and survival.

DETAILED DESCRIPTION:
The complex intervention in AlloLife will consist of a set of technically-supported tools that will enable active care management through the patient and treating physician to improve QoL.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patients with performed allogeneic stem cell transplantation any type of donor, stem cell source, GVHD prophylaxis or conditioning regimen and at least at day +20 after HCT.
* Hematologic Remission after HCT at study entrance, MRD positive patients are allowed to enter the study
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Signature of informed and written consent by the subject or by the subject's legally acceptable representative for patients under guardianship or trusteeship to participate in the study
* Access to an internet connected device (smartphone/tablet/computer)
* Able to understand and communicate in the respective language
* Consent to use a wearable device through the time of the study
* Consent to use a chatbot application for both healthcare data exchange and psychologic intervention

Exclusion Criteria:

* Missing consent to use a wearable device and contribute personal data collected at the point of life to the study
* ECOG performance status of 4
* Relapse of the disease at study inclusion
* Uncontrolled systemic infection
* Diagnosis of a secondary malignancy requiring systemic therapy
* Reported ongoing severe depression or potential suicidal ideation
* Vulnerable patients such as: minor, persons deprived of liberty, persons in Intensive Care Unit unable to provided informed consent prior to the intervention
* Other ongoing interventional protocol that might interfere with the current study primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life as measured by the FACT-BMT score | 12 months
  Change in QoL measured by the FACT BMT score on a continuous scale. The Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) as initially developed by McQuellon RP et al. BMT 1997. It scales between 0 (zero) and 196 on a continuous scale, where higher values refer to higher Quality of Life.

IPD SHARING:
Plan to Share IPD: Undecided
The IPD Sharing Plan will be developed during the project.